CLINICAL TRIAL: NCT04499729
Title: Implementing IntelliCare in Collaborative Care: A Quality Improvement Evaluation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment site (Rush University Medical Center Collaborative Care Program) redefined their service objectives such that IntelliCare was no longer a good fit.
Sponsor: Adaptive Health, Inc (Industry)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R44MH114725 (NIH)
Record Dates: First submitted 2020-07-27; First posted 2020-08-05 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: We will utilize a pragmatic, system-wide rollout quality improvement evaluation design. Data from patients in the Rush Collaborative Care service will be used beginning Dec 1, 2019. The first care manager will begin offering IntelliCare as part of the collaborative care service in September, 2020, and one additional care manager will begin offering IntelliCare to patients every 3 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): TAU will be the treatment that is provided through the Rush Collaborative Care program as part of their service
  Interventions: Behavioral: Treatment as Usual (TAU)
- IntelliCare (Experimental): Patients will be offered IntelliCare as part of their care in the Rush Collaborative Care service. Patients who agree will download the IntelliCare app, which provides self management and collects symptom self-report data. Symptom severity scores are displayed to the care manager, allowing them to manage the patient's care. The app also provides a secure messaging service for communication between the care manager and the patient.
  Interventions: Device: IntelliCare

INTERVENTIONS:
Device: IntelliCare — IntelliCare provides self management and collects symptom self-report data. Symptom severity scores are displayed to the care manager, allowing them to manage the patient's care. The app also provides a secure messaging service for communication between the care manager and the patient.
  Arms: IntelliCare
Behavioral: Treatment as Usual (TAU) — Treatment as usual in the Rush Collaborative Care service
  Arms: Treatment as Usual (TAU)

SUMMARY:
The overarching aim of the proposed project is to conduct a pragmatic, quality improvement evaluation of the IntelliCare Platform for improving processes of care in the Rush Collaborative Care program, and improving patient population depression outcomes, to determine the long-term utility of IntelliCare for Rush.

DETAILED DESCRIPTION:
This study is a pragmatic, system-wide rollout quality improvement evaluation design displayed in Figure 1. The Rush IRB has waived consent for this quality improvement trial. Data from the EHR will be used beginning December 1, 2019. The first care manager (CM) will begin enrolling patients into IntelliCare in September, 2020. Additional CMs will begin using IntelliCare at approximately 3 month intervals. In September 2021, support for IntelliCare from the evaluation team will be withdrawn, to examine the sustainability of the IntelliCare Platform.

Patients Data from all patients, aged 18 or older, enrolled collaborative care from December 1, 2019 through August 31, 2022 will be used to evaluate the IntelliCare service. All CCT patients who are 18 or older, and have a smartphone will be offered enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Rush Collaborative Care service
* Owns a personal smartphone

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Depression | Up to 20 Months
  Patient Health Questionnaire-9 (PHQ-9) assessment for depression
Number of assessments | Up to 20 Months
  Number of Patient Health Questionnaire (PHQ-9) assessments acquired in the EHR

SECONDARY OUTCOMES:
First to last assessment | Up to 20 Months
  Time from first to last PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn MacIver, Principal Investigator — Adaptive Health
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is not current plan to share IPD outside the research team.